CLINICAL TRIAL: NCT01603628
Title: BOTOX® Treatment in Pediatric Lower Limb Spasticity: Double-blind Study
Brief Title: BOTOX® Treatment in Pediatric Lower Limb Spasticity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 191622-111; 2012-000042-35 (EudraCT Number)
Record Dates: First submitted 2012-05-21; First posted 2012-05-22 (Estimated); Results first posted 2018-08-14 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-07

CONDITIONS: Pediatrics; Muscle Spasticity; Cerebral Palsy
MeSH Terms: conditions — Muscle Spasticity; Cerebral Palsy | interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- BOTOX® 4 U/kg (Experimental): Participants received intramuscular injections of BOTOX® (botulinum toxin Type A) 4 U per kg of body weight (4 U/kg) into specified muscles of the lower limb on Day 1. Participants received weekly physical therapy (PT).
  Interventions: Biological: botulinum toxin Type A
- BOTOX® 8 U/kg (Experimental): Participants received intramuscular injections of BOTOX® (botulinum toxin Type A) 8 U per kg of body weight (8 U/kg) into specified muscles of the lower limb on Day 1. Participants received weekly PT.
  Interventions: Biological: botulinum toxin Type A
- Normal Saline (Placebo) (Placebo Comparator): Participants received intramuscular injections of normal saline (placebo) into specified muscles of the lower limb on Day 1. Participants received weekly PT.
  Interventions: Drug: Normal Saline (Placebo)

INTERVENTIONS:
Biological: botulinum toxin Type A — Participants received intramuscular injections of botulinum toxin Type A into specified muscles of the lower limb on Day 1.
  Other Names: BOTOX®
  Arms: BOTOX® 4 U/kg; BOTOX® 8 U/kg
Drug: Normal Saline (Placebo) — Participants received intramuscular injections of normal saline (placebo) into specified muscles of the lower limb on Day 1.
  Arms: Normal Saline (Placebo)

SUMMARY:
This study will evaluate the safety and efficacy of BOTOX® (botulinum toxin Type A) in pediatric patients with lower limb spasticity.

ELIGIBILITY:
Inclusion Criteria:

* Minimum weight of 10 kg/22 lb
* Cerebral palsy with dynamic muscle contracture /spasticity of the ankle

Exclusion Criteria:

* Muscular dystrophy, myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, or mitochondrial disease
* Uncontrolled epilepsy
* Botulinum Toxin therapy of any serotype for any condition within the last 6 months
* History of surgical intervention of the lower study leg or planned surgery of any limb during the study
* Previous casting of the study limb for spasticity within 6 months or with a dynamic splint within 3 months, or planned casting or dynamic splinting for spasticity of the study limb or affected upper limb during the study

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 384 (Actual)
Dates: Start 2012-09-11 (Actual); Primary Completion 2017-06-28 (Actual); Study Completion 2017-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rozalina Dimitrova, Study Director — Allergan
Locations (53):
- United States (24):
  - AMS Neurology, Pasadena, California
  - Harrison Clinical Management, Pomona, California
  - Children's Hospital Colorado Dept. of PM&R, Aurora, Colorado
  - Associated Neurologists of Southern CT, P.C., Fairfield, Connecticut
  - New England Center for Clinical Research, Stamford, Connecticut
  - NW FL Clinical Research Group, LLC, Gulf Breeze, Florida
  - Axcess Medical Research, LLC, Loxahatchee Groves, Florida
  - Pediatric Neurology, PA, Orlando, Florida
  - Children's Healthcare of Atlanta Children's Rehabilitation Associates, Atlanta, Georgia
  - Rehab Institute of Chicago, Chicago, Illinois
  - The Children's Mercy Hospital & Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Clinical Research Center of New Jersey, Voorhees Township, New Jersey
  - NYU Hospital for Joint Diseases, New York, New York
  - Columbia University Medical Center Dept. of Rehab. & Regenerative Medicine, New York, New York
  - OnSite Clinical Solutions, LLC, Charlotte, North Carolina
  - PMG Research of Charlotte, LLC, Charlotte, North Carolina
  - Rhode Island Hospital, Providence, Rhode Island
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine Texas Children's Hospital, Houston, Texas
  - Road Runner Research, San Antonio, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - Marshfield Clinic, Marshfield, Wisconsin
- Hungary (2):
  - Semmelweis Egyetem- Ortopédiai Klinika, Budapest
  - Debrecen University Clinical Center, Orthopedic Clinic, Debrecen
- Istituto IRCCS G. Gaslini, Genoa, Italy
- Philippines (3):
  - Philippine Orthopedic Center, Quezon City
  - St. Luke's Medical Center-Quezon City, Quezon City
  - Philippine Children's Medical Center, Quezon City
- Poland (9):
  - Uniwersytecki Dzieciecy Szpita, Bialystok
  - Uni Centrum Kliniczne, Gdansk
  - Centrum Rehabilitacji Krok po Kroku, Gdansk
  - Specjal. Gabinet Neurologiczny, Krakow
  - INTERMED, Lublin, Lublin
  - CRH ŻAGIEL MED, Lublin, Lublin
  - Szpital Wojewódzki Nr 2, Rzeszów
  - Neuro - Dzieci I Mlodziezy Aga, Warsaw
  - NZOZ Mazowieckie Centrum, Warsaw
- Russia (3):
  - Childrens Republic Hospital, Kazan'
  - Smolensk Regional Hospital- Regional Budget State Healthcare institution, Smolensk
  - Tyumen Regional Hospital #2 - State Budget Healthcare Institution of Tyumen region, Tyumen
- South Korea (6):
  - Daegu Fatima Hospital, Daegu
  - National Health Insurance Service Ilsan Hospital, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
- Thailand (2):
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai University, Chiang Mai
  - Srinagarind Hospital, Khon Kaen University, Khon Kaen
- Turkey (Türkiye) (3):
  - Ankara Diskapi Yildrim Beyazit, Ankara
  - Kocaeli Üniversitesi, Kocaeli
  - Selçuk Üniversitesi, Konya

REFERENCES:
- See also: Additional information on study locations near you may be found at AllerganClinicalTrials.com. For any study not on AllerganClinicalTrials.com, please contact IR-CTRegistration@Allergan.com for assistance. — http://www.allerganclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Pediatric participants with lower limb spasticity were randomized 1:1:1 to one of three treatment groups: BOTOX® 4 or 8 U/kg (unit per kilogram) or placebo.
Groups:
- BOTOX® 8 U/kg: Participants received intramuscular injections of BOTOX® (botulinum toxin Type A) 8 units (U) per kg of body weight (8 U/kg) into specified muscles of the lower limb on Day 1. Participants received weekly physical therapy (PT).
- BOTOX® 4 U/kg: Participants received intramuscular injections of BOTOX® (botulinum toxin Type A) 4 U per kg of body weight (4 U/kg) into specified muscles of the lower limb on Day 1. Participants received weekly PT.
- Placebo: Participants received intramuscular injections of normal saline (placebo) into specified muscles of the lower limb. Participants received weekly PT.
Period: Overall Study
Arm/Group | BOTOX® 8 U/kg | BOTOX® 4 U/kg | Placebo
Started | 128 | 126 | 130
Safety Population: Received Treatment | 128 | 126 | 128
Completed | 125 | 123 | 128
Not Completed | 3 | 3 | 2
Not completed — Personal Reasons | 1 | 1 | 2
Not completed — Protocol Violation | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Other Miscellaneous Reason | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- BOTOX® 8 U/kg: Participants received intramuscular injections of BOTOX® (botulinum toxin Type A) 8 U per kg of body weight (8 U/kg) into specified muscles of the lower limb on Day 1. Participants received weekly physical therapy (PT).
- Total: Total of all reporting groups
Arm/Group | BOTOX® 8 U/kg | BOTOX® 4 U/kg | Placebo | Total
Number analyzed (Participants) | 128 | 126 | 130 | 384
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.7 (3.90) | 6.4 (3.58) | 6.6 (3.89) | 6.6 (3.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 58 | 62 | 177
  Male | 71 | 68 | 68 | 207
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 77 | 76 | 80 | 233
  Black | 2 | 3 | 4 | 9
  Asian | 42 | 35 | 38 | 115
  Hispanic | 7 | 10 | 6 | 23
  Other Not Specified | 0 | 1 | 3 | 4
Modified Ashworth Scale-Bohannon (MAS-B) Ankle Score with Knee Extended [Mean (Standard Deviation); unit: score on a scale] — The MAS-B evaluates spasticity, grading the resistance encountered in the principal muscle group (elbow and wrist) by passively moving a limb through its range of motion at a specified velocity. The resistance encountered to passive stretch was graded on a 6-point scale: 0=no increase in muscle tone (best) to 4=affected part(s) rigid in flexion or extension (worst). For analysis purposes, the MAS-B was recoded as follows: 0=1, 1=1, 1+=2, 2=3, 3=4, 4=5. Population: 2 participants in the Placebo arm are not included in the analysis.
  score on a scale
    number analyzed (Participants) | 128 | 126 | 128 | 382
    (all) | 3.5 (0.52) | 3.5 (0.53) | 3.5 (0.50) | 3.5 (0.52)

OUTCOME MEASURES:

1. Primary Outcome: Average Change From Baseline in Modified Ashworth Scale-Bohannon (MAS-B) Ankle Score With Knee Extended at Weeks 4 and 6
Description: The MAS-B was used to evaluate spasticity based on grading the resistance encountered in the principal muscle group (elbow and wrist) by means of passively moving a limb through its range of motion at a study specified velocity. The resistance encountered to passive stretch was graded using a 6-point scale where: 0=no increase in muscle tone (best) to 4=affected part(s) rigid in flexion or extension (worst). For analysis purposes, the MAS-B was recoded as follows: 0=1, 1=1, 1+=2, 2=3, 3=4, 4=5. The scores at Weeks 4 and 6 were averaged. A Mixed Model Repeated Measures (MMRM) model was used for analysis. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 1) to Weeks 4 and 6
Population: Participants from the mITT population, all randomized participants with a valid MAS-B baseline ankle score with knee extended and at least one post-baseline measurement at Weeks 2, 4, or 6 for the MAS-B of the ankle score with knee extended and the CGI by physician, with data available for analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | BOTOX® 8 U/kg | BOTOX® 4 U/kg | Placebo
Number analyzed (Participants) | 123 | 119 | 125
score on a scale | -1.06 (0.071) | -1.01 (0.072) | -0.80 (0.071)
Statistical Analysis 1: Comparison: BOTOX® 8 U/kg vs Placebo; Test type: Superiority; p = 0.010, Mixed Model Repeated Measures — MMRM including baseline MAS-B ankle score (knee extended) as a covariate and factors of age, treatment, visit, treatment-by-visit interaction, study center and previous botulinum toxin exposure where age is represented by stratification categories; Least Squares (LS) Mean Difference = -0.26, 95% CI 2-sided [-0.453 to -0.063]
Statistical Analysis 2: Comparison: BOTOX® 4 U/kg vs Placebo; Test type: Superiority; p = 0.033, Mixed Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -0.21, 95% CI 2-sided [-0.405 to -0.018]

2. Primary Outcome: Average Clinical Global Impression (CGI) of Overall Change by Physician at Weeks 4 and 6
Description: The CGI of overall change (improvement or worsening) was assessed by the physician considering the participant's clinical condition and severity of side effects using a 9-point scale where: -4=very marked worsening to +4=very marked improvement. The scores at Weeks 4 and 6 were averaged. A Mixed Model Repeated Measures (MMRM) model was used for analysis.
Time Frame: Weeks 4 and 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | BOTOX® 8 U/kg | BOTOX® 4 U/kg | Placebo
Number analyzed (Participants) | 123 | 118 | 124
score on a scale | 1.65 (0.090) | 1.49 (0.091) | 1.36 (0.089)
Statistical Analysis 1: Comparison: BOTOX® 8 U/kg vs Placebo; Test type: Superiority; p = 0.023, Mixed Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = 0.29, 95% CI 2-sided [0.040 to 0.532]
Statistical Analysis 2: Comparison: BOTOX® 4 U/kg vs Placebo; Test type: Superiority; p = 0.299, Mixed Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = 0.13, 95% CI 2-sided [-0.115 to 0.374]

3. Secondary Outcome: Goal Attainment Score (GAS) as Assessed by Physician Using a 6-Point Scale
Description: Two functional goals, one active and one passive, were selected by the participant and family in consultation with the physician investigator and/or treating physical therapist relative to the lower limb impairment due to spasticity. The physician assessed the achievement of the goals using a 6-point scale: where -3=worse than start to +2=much more than expected: improvements clearly exceed the defined therapeutic goal. An Analysis of Covariance (ANCOVA) model was used for analysis.
Time Frame: Weeks 8 and 12
Population: Participants from the mITT population, all randomized participants with a valid MAS-B baseline ankle score with knee extended and at least one post-baseline measurement at Weeks 2, 4, or 6 for the MAS-B of the ankle score with knee extended and the CGI by physician, with data available for analysis at the given time-point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | BOTOX® 8 U/kg | BOTOX® 4 U/kg | Placebo
Number analyzed (Participants) | 127 | 125 | 129
score on a scale
  Week 8, Active Goal: number analyzed (Participants) | 121 | 121 | 127
  Week 8, Active Goal | 0.10 (0.108) | -0.03 (0.108) | -0.31 (0.105)
  Week 8, Passive Goal: number analyzed (Participants) | 120 | 121 | 127
  Week 8, Passive Goal | 0.19 (0.115) | 0.18 (0.114) | -0.26 (0.111)
  Week 12, Active Goal: number analyzed (Participants) | 124 | 123 | 128
  Week 12, Active Goal | 0.37 (0.112) | 0.09 (0.113) | -0.12 (0.111)
  Week 12, Passive Goal: number analyzed (Participants) | 124 | 123 | 128
  Week 12, Passive Goal | 0.40 (0.114) | 0.27 (0.114) | 0.00 (0.112)
Statistical Analysis 1: Comparison: BOTOX® 8 U/kg vs Placebo; Week 8, Active Goal; Test type: Superiority; p = 0.005, ANCOVA — ANCOVA model including baseline MAS-B ankle score with knee extended as a covariate and factors of age group, treatment group, study center and previous botulinum toxin exposure where age group is represented by stratification categories; LS Mean Difference = 0.41, 95% CI 2-sided [0.126 to 0.704]
Statistical Analysis 2: Comparison: BOTOX® 4 U/kg vs Placebo; Week 8, Active Goal; Test type: Superiority; p = 0.047, ANCOVA — [p-value comment as in outcome 3, analysis 1]; LS Mean Difference = 0.29, 95% CI 2-sided [0.004 to 0.573]
Statistical Analysis 3: Comparison: BOTOX® 8 U/kg vs Placebo; Week 8, Passive Goal; Test type: Superiority; p = 0.004, ANCOVA — [p-value comment as in outcome 3, analysis 1]; LS Mean Difference = 0.45, 95% CI 2-sided [0.145 to 0.756]
Statistical Analysis 4: Comparison: BOTOX® 4 U/kg vs Placebo; Week 8, Passive Goal; Test type: Superiority; p = 0.004, ANCOVA — [p-value comment as in outcome 3, analysis 1]; LS Mean Difference = 0.44, 95% CI 2-sided [0.141 to 0.740]
Statistical Analysis 5: Comparison: BOTOX® 8 U/kg vs Placebo; Week 12, Active Goal; Test type: Superiority; p = 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; LS Mean Difference = 0.49, 95% CI 2-sided [0.191 to 0.797]
Statistical Analysis 6: Comparison: BOTOX® 4 U/kg vs Placebo; Week 12, Active Goal; Test type: Superiority; p = 0.153, ANCOVA — [p-value comment as in outcome 3, analysis 1]; LS Mean Difference = 0.22, 95% CI 2-sided [-0.081 to 0.541]
Statistical Analysis 7: Comparison: BOTOX® 8 U/kg vs Placebo; Week 12, Passive Goal; Test type: Superiority; p = 0.010, ANCOVA — [p-value comment as in outcome 3, analysis 1]; LS Mean Difference = 0.41, 95% CI 2-sided [0.100 to 0.711]
Statistical Analysis 8: Comparison: BOTOX® 4 U/kg vs Placebo; Week 12, Passive Goal; Test type: Superiority; p = 0.078, ANCOVA — [p-value comment as in outcome 3, analysis 1]; LS Mean Difference = 0.27, 95% CI 2-sided [-0.031 to 0.571]

4. Secondary Outcome: Change From Baseline in Severity of Spasticity of the Ankle With Knee Extended and Knee Flexed (R2-R1) Calculated Using the Modified Tardieu Scale (MTS)
Description: The MTS measured the difference between slow and fast range of motion (R2-R1) and respective change from baseline to each posttreatment office visit. The MTS of the ankle was used to determine the passive range of movement at different movement velocities, V1 (as slow as possible) and V3 (as fast as possible) with the relative difference between a slow and fast velocity passive stretch determining the dynamic component of the muscle contracture for the joint. The investigator measured 2 joint angles by goniometer: the R1 angle which is the angle of catch after a fast velocity (V3) stretch and the R2 angle defined as the passive joint range of movement following a slow velocity (V1) stretch. The R2-R1 value indicated the level of the dynamic component of spasticity in the joint. The difference between R2 and R1 range of motion and respective change from baseline to each posttreatment office visit on the MTS was derived. An Analysis of Covariance (ANCOVA) model was used for analysis.
Time Frame: Baseline (Day 1) to Weeks 2, 4, 6, 8 and 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: degrees
Arm/Group | BOTOX® 8 U/kg | BOTOX® 4 U/kg | Placebo
Number analyzed (Participants) | 127 | 125 | 129
degrees
  Change from Baseline to Week 2: number analyzed (Participants) | 126 | 124 | 129
  Change from Baseline to Week 2 | -4.44 (1.023) | -5.69 (1.024) | -2.44 (1.0101)
  Change from Baseline to Week 4: number analyzed (Participants) | 124 | 121 | 126
  Change from Baseline to Week 4 | -6.11 (1.134) | -6.80 (1.135) | -4.69 (1.121)
  Change from Baseline to Week 6: number analyzed (Participants) | 126 | 121 | 126
  Change from Baseline to Week 6 | -6.65 (1.029) | -7.23 (1.049) | -3.32 (1.029)
  Change from Baseline to Week 8: number analyzed (Participants) | 122 | 123 | 127
  Change from Baseline to Week 8 | -5.42 (1.317) | -5.82 (1.308) | -3.36 (1.291)
  Change from Baseline to Week 12: number analyzed (Participants) | 125 | 123 | 128
  Change from Baseline to Week 12 | -4.59 (1.070) | -3.07 (1.074) | -1.98 (1.057)
Statistical Analysis 1: Comparison: BOTOX® 8 U/kg vs Placebo; Change from Baseline to Week 2; Test type: Superiority; p = 0.158, ANCOVA — ANCOVA model including baseline MTS ankle score with knee extended as a covariate and factors of age group, treatment group, study center, and previous botulinum toxin exposure where age group is represented by stratification categories; LS Mean Difference = -1.99, 95% CI 2-sided [-4.768 to 0.779]
Statistical Analysis 2: Comparison: BOTOX® 4 U/kg vs Placebo; Change from Baseline to Week 2; Test type: Superiority; p = 0.020, ANCOVA — [p-value comment as in outcome 4, analysis 1]; LS Mean Difference = -3.25, 95% CI 2-sided [-5.974 to -0.524]
Statistical Analysis 3: Comparison: BOTOX® 8 U/kg vs Placebo; Change from Baseline to Week 4; Test type: Superiority; p = 0.363, ANCOVA — [p-value comment as in outcome 4, analysis 1]; LS Mean Difference = -1.42, 95% CI 2-sided [-4.489 to 1.648]
Statistical Analysis 4: Comparison: BOTOX® 4 U/kg vs Placebo; Change from Baseline to Week 4; Test type: Superiority; p = 0.171, ANCOVA — [p-value comment as in outcome 4, analysis 1]; LS Mean Difference = -2.11, 95% CI 2-sided [-5.127 to 0.914]
Statistical Analysis 5: Comparison: BOTOX® 8 U/kg vs Placebo; Change from Baseline to Week 6; Test type: Superiority; p = 0.020, ANCOVA — [p-value comment as in outcome 4, analysis 1]; LS Mean Difference = -3.33, 95% CI 2-sided [-6.143 to -0.525]
Statistical Analysis 6: Comparison: BOTOX® 4 U/kg vs Placebo; Change from Baseline to Week 6; Test type: Superiority; p = 0.006, ANCOVA — [p-value comment as in outcome 4, analysis 1]; LS Mean Difference = -3.92, 95% CI 2-sided [-6.688 to -1.148]
Statistical Analysis 7: Comparison: BOTOX® 8 U/kg vs Placebo; Change from Baseline to Week 8; Test type: Superiority; p = 0.254, ANCOVA — [p-value comment as in outcome 4, analysis 1]; LS Mean Difference = -2.07, 95% CI 2-sided [-5.621 to 1.491]
Statistical Analysis 8: Comparison: BOTOX® 4 U/kg vs Placebo; Change from Baseline to Week 8; Test type: Superiority; p = 0.165, ANCOVA — [p-value comment as in outcome 4, analysis 1]; LS Mean Difference = -2.46, 95% CI 2-sided [-5.935 to 1.014]
Statistical Analysis 9: Comparison: BOTOX® 8 U/kg vs Placebo; Change from Baseline to Week 12; Test type: Superiority; p = 0.078, ANCOVA — [p-value comment as in outcome 4, analysis 1]; LS Mean Difference = -2.61, 95% CI 2-sided [-5.517 to 0.296]
Statistical Analysis 10: Comparison: BOTOX® 4 U/kg vs Placebo; Change from Baseline to Week 12; Test type: Superiority; p = 0.451, ANCOVA — [p-value comment as in outcome 4, analysis 1]; LS Mean Difference = -1.09, 95% CI 2-sided [-3.944 to 1.758]

ADVERSE EVENTS:
Time Frame: Baseline (Day 1) to the end of study (Week 12)
Description: The Safety Population, all treated participants based on the treatment received, was used to determine the number of participants at risk for Serious Adverse Events and Adverse Events.
Arm/Group | BOTOX® 8 U/kg | BOTOX® 4 U/kg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/128 | 0/126 | 0/128
Serious Adverse Events (participants affected / at risk) | 0/128 | 3/126 | 4/128
Other Adverse Events (participants affected / at risk) | 24/128 | 26/126 | 35/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BOTOX® 8 U/kg (N=128) | BOTOX® 4 U/kg (N=126) | Placebo (N=128)
Extrasystoles (Cardiac disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Gastoeneteritis (Infections and infestations) | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 1 | 2
Radicular Pain (Nervous system disorders) | 0 | 0 | 1
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BOTOX® 8 U/kg (N=128) | BOTOX® 4 U/kg (N=126) | Placebo (N=128)
Pyrexia (General disorders) | 5 | 8 | 7
Viral upper respiratory tract infection (Infections and infestations) | 12 | 14 | 22
Upper respiratory tract infection (Infections and infestations) | 8 | 10 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-08-16): https://cdn.clinicaltrials.gov/large-docs/28/NCT01603628/SAP_000.pdf
  • Study Protocol (2016-07-25): https://cdn.clinicaltrials.gov/large-docs/28/NCT01603628/Prot_001.pdf